CLINICAL TRIAL: NCT05759091
Title: The Effect of Applying Cognitive Defusion Techniques on Mindful Awareness, Cognitive Fusion and Believability of Delusions Among Clients With Schizophrenia: A Randomized Control Trial
Brief Title: Effect of Applying Cognitive Defusion Techniques on Mindful Awareness, Cognitive Fusion and Believability of Delusions Among Clients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, ayman el-ashry, lecturer of psychiatric nursing and mental health department, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00013620/63/9/2022
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia; Psychosis; Nurse's Role; Delusions
Keywords: Believability of Delusions; Cognitive Defusion techniques; Cognitive Fusion; Mindful Awareness; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Delusions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive defusion interventional group (Experimental): patients with schizophrenia who suffer from persistent delusions participated in cognitive defusion techniques on individual base through sex sessions twice weekly with homework assignments between sessions and skills demonstration by simulation and psychodrama.
  Interventions: Behavioral: cognitive defusion techniques
- control group (No Intervention): patients with schizophrenia who suffer from persistent delusions participated in usual routine care in the hospital.

INTERVENTIONS:
Behavioral: cognitive defusion techniques — Defusing from your delusions helps to lessen their negative impact on your behaviour. So defusion is a vital step towards being able to act flexibly, in accordance with core values, instead of being dictated to by inflexible rules, reasons, judgments etc. There are numerous exercises in ACT Companion with a focus on identifying unhelpful thoughts which would benefit from defusion, or building defusion skills, most of which are found in the open up section of the app. Some of these are reading and writing exercises, and some are guided meditation audio recordings.
  ACT Companion defusion exercises
  1. Letting go
  2. Not good enough
  3. Thought defusion
  4. Observing your thoughts
  5. Labelling thoughts and feelings
  6. I am having the thought that.....
  7. milk.milk.milk exercise
  8. silly voice exercise, passenger on the bus, tug of war with a monster
  Arms: cognitive defusion interventional group

SUMMARY:
Schizophrenia causes hallucinations, delusions, and disorganized thinking, resulting in decreased functioning and lifelong therapy.Delusion believability is the degree of belief in the truth of one's subjective experiences as representations of reality. It was unpleasant, typically accompanied by a suspicious, strange tension. Delusional belief is seen as a means of resolving tension and conflict in cognition and experience. Previous studies have shown that cognitive defusion strategies help people become more aware of their surroundings, accept their thoughts and feelings, and become more psychologically adjustable. defusion is crucial in reducing medication-resistant psychotic symptoms such delusions in schizophrenia patients. Therefore, this study aimed to investigate the effects of cognitive defusion techniques on psychological flexibility, mindful awareness, cognitive fusion, and believability of delusions among clients with schizophrenia.

Research Hypothesizes

* Clients who participated in cognitive defusion techniques had more psychological flexibility and mindful awareness than the control group.
* Clients who participated in cognitive defusion techniques had less cognitive fusion and delusional believability than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Male clients diagnosed with schizophrenia according to the DSM-V
* Diagnosed with schizophrenia With no comorbidity.
* Able to communicate coherently and relevantly.
* Able to read and write.
* Willing to participate in the study
* Duration of illness not exceeding 10 years.

Exclusion Criteria:

• Any client in an acute phase or have any neurological disorder that may affect cognitive function were excluded from a study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only male patients with schizophrenia included in this study to decrease confounding factors.
Enrollment: 70 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
The Acceptance and Action Questionnaire-II (AAQII) | up to 14 weeks
  It is a seven-item self-reported scale developed to measure of psychological flexibility, with items targeted to several of the six key processes: defusion, acceptance, and committed action (example item: 'I worry about not being able to control my worries and feelings'.). Each item is followed by a seven-category response scale, started from never true (1), very seldom true (2), seldom true (3), sometimes true (4), frequently true (5), almost always true (6) to always true (7). Higher scores indicate greater psychological inflexibility (total score range: 7-49, calculated as the sum of the item responses). Previous research has reported a Cronbach's of 0.84.
The Cognitive Fusion Questionnaire-7 (CFQ-7) | up to 14 weeks
  It is designed to elicit one's level of cognitive fusion (example item: 'I find it easy to view my thoughts from a different perspective'.). Respondents rate each of 7 items on a 7- Likert scale ranging from 1 'Never true' to 7 'Always true'. Higher scores on the CFQ indicate greater cognitive fusion (total score range: 7-49, calculated as a sum of the responses). Studies demonstrate satisfactory reliability with a Cronbach's of 0.86.
Southampton Mindfulness Questionnaire (SMQ) | up to 14 weeks
  Southampton Mindfulness Questionnaire is a 16-item scale that assesses the relationship one establishes with distressing thoughts and images (e.g., "I am able just to notice them without reacting"). Items are scored on a 7-point Likert scale, ranging from strongly disagree (0) to strongly agree (6). In the original study, the Cronbach's alpha obtained was 0.89.
Psychotic Symptom Rating Scales (PSYRATS-D) | up to 14 weeks
  It consists of 17 items divided into two subscales designed to rate auditory hallucinations and delusions. In this study, only the delusion subscale (PSYRATS-D) was used. The Delusion subscale measures various dimensions of delusion through 6 items divided into emotional characteristics (distress) and cognitive interpretation subscales. The first subscale is for cognitive interpretation (4 items) includes Amount of preoccupation with delusions, Duration of preoccupation with delusions, Conviction, and Disruption to life caused by beliefs. The second subscale is for emotional distress of delusions (2 items) Amount of Distress, and Intensity of Distress. The PSYRATS-AH was rated on a five-point Likert scale ranging from 0 (not endorsing the item) to 4 (fully endorsing the item). With a total score range from 0 to 24. The PSYRATS-D has been found to have high inter-rater reliability (0.99-1) and test-retest reliability (r = 0.70).

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Mohamed El-Ashry, PHD, Principal Investigator — Faculty of nursing, Alexandria University, Egypt
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bach P, Hayes SC. The use of acceptance and commitment therapy to prevent the rehospitalization of psychotic patients: a randomized controlled trial. J Consult Clin Psychol. 2002 Oct;70(5):1129-39. doi: 10.1037//0022-006x.70.5.1129. PMID 12362963
- [Background] Hayes SC. Acceptance and Commitment Therapy, Relational Frame Theory, and the Third Wave of Behavioral and Cognitive Therapies - Republished Article. Behav Ther. 2016 Nov;47(6):869-885. doi: 10.1016/j.beth.2016.11.006. Epub 2016 Nov 10. PMID 27993338
- [Background] Boge K, Pollex F, Bergmann N, Hahne I, Zierhut MM, Mavituna S, Thomas N, Hahn E. Mindfulness, cognitive fusion, and self-compassion in patients with schizophrenia spectrum disorders-A cross-sectional study. Front Psychiatry. 2022 Aug 2;13:959467. doi: 10.3389/fpsyt.2022.959467. eCollection 2022. PMID 35982935
- [Derived] El-Ashry AM, Abd Elhay ES, Taha SM, Khedr MA, Attalla Mansour FS, Alabdullah AAS, Farghaly Abdelaliem SM, El-Sayed MM. Effect of applying nursing-based cognitive defusion techniques on mindful awareness, cognitive fusion, and believability of delusions among clients with schizophrenia: a randomized control trial. Front Psychiatry. 2024 Apr 26;15:1369160. doi: 10.3389/fpsyt.2024.1369160. eCollection 2024. PMID 38736628